CLINICAL TRIAL: NCT03759899
Title: Establishment of Clinical Applicable Human Amniotic Epithelial Cell Products and Its Preliminary Application in Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: hAECs Are Preliminarily Applied in Allogeneic Hematopoietic Stem Cell Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director of the Hematology Department, Peking University People's Hospital
Other Study IDs: 2018PHB007-01
Record Dates: First submitted 2018-11-19; First posted 2018-11-30 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
hAECs Are Preliminarily Applied in Allogeneic Hematopoietic Stem Cell Transplantation

DETAILED DESCRIPTION:
Establishment of Clinical Applicable Human Amniotic Epithelial Cell Products and Its Preliminary Application in Allogeneic Hematopoietic Stem Cell Transplantation

ELIGIBILITY:
Inclusion Criteria:

* leukemia patients with allogeneic HSCT
* KFS score >90
* after transplantation, the patient was implanted (peripheral blood neutrophil absolute value >500/ul for 3 consecutive days)
* no uncontrolled infection after transplantation
* activity II above aGVHD
* patients agreed to participate in the study

Exclusion Criteria:

* patients refused to participate in the study
* patients have poor compliance
* has received hormone therapy
* patients had serious heart, lung, liver, kidney and other vital organs damage
* researchers believe that patients who are not suitable for observation study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: leukemia patients with allogeneic HSCT
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Cell counts of T cells, NK cells, B cells and monocytes | Day 7
  proliferation and apoptosis of T cells, NK cells, B cells and monocytes in peripheral blood of patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided